CLINICAL TRIAL: NCT05462015
Title: Effects of Elastic Band Resistance Training on Physical Fitness and Risk of Falls in Old Adults With Hospitalized and High Fall Risk.
Brief Title: Elastic Band Resistance Training on Physical Fitness and Risk of Falls in Elderly.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulty in hospital caused by COVID-19
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Gong-Hong Lin, Assistant Professor, Taipei Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202205064
Record Dates: First submitted 2022-07-11; First posted 2022-07-18 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Falls; Old Age; Debility; Hospitalisation; Resistance Training; Physical Fitness
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic band (Experimental): The experimental group received a 35-minute training course for 2 weeks, 3 times a week, each time during the hospitalization. A total of 4 assessments were performed: baseline (pre-intervention), after third-time intervention, post-intervention, and one week after the intervention.
  Interventions: Behavioral: elastic-band exercises
- Control (Active Comparator): The control group was given routine rehabilitation exercise
  Interventions: Behavioral: regular rehabilitation

INTERVENTIONS:
Behavioral: elastic-band exercises — The training content includes 5 minutes of warm-up exercise, 20 minutes of elastic-band resistance training, and 10 minutes of cool-down exercise.
  Other Names: resistance band exercises
  Arms: Elastic band
Behavioral: regular rehabilitation — The training content includes 5-minute warm-up exercise, 20-minute upper and lower extremity muscle strengthening, and 10-minute cool-down exercise
  Arms: Control

SUMMARY:
A lack of studies has applied elastic band resistance training exercises on hospitalized elderly, so the effect of elastic band resistance training exercises on physical fitness and risk of falls was unclear. Therefore, the purposes of this study were to investigate the effectiveness of elastic band resistance training on improving physical fitness and reducing the risk of falls in hospitalized elderly with high risk of falls. This study is an experimental study. The experimental group was given 3 times a week for 2 consecutive weeks of elastic band resistance training, while the control group was given regular rehabilitation exercises. The differences in physical fitness and fall risk between the two groups were examined.

ELIGIBILITY:
Inclusion Criteria:

1. Elders are over 65 years old and admitted to this medical ward due to acute/chronic disease
2. Elders have no physical impairment
3. Elders have a clear cognition, can follow movement commands in Chinese or Taiwanese
4. Elders have greater than 4 points in lower extremity muscle strength measured by the Manual Muscle Power Test
5. Elders have greater than 45 points in the Morse Fall Scale, which indicate a high risk of falling

Exclusion Criteria:

1. Unclear consciousness
2. Unable to follow the execution of elastic band resistance training
3. With restricted activities, musculoskeletal disorders, or nerve diseases
4. Unsuitable athletic trainers

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Functional Fitness Test | first day
  Physical fitness is considered to be the comprehensive ability of the body to adapt to life and the environment; people with good physical fitness have good vitality and adaptability in daily life or work, physical activities or sports, and are not prone to fatigue or weakness; Ministry of Health and Welfare National Health Administration refers to the United States Scholars have designed functional fitness tests for the elderly over 60 years old, and developed domestic fitness tests to assess physical health. Topics include muscle strength and endurance, cardiorespiratory endurance, flexibility, agility, and homeostasis. Scholars in Taiwan conducted a reliability and validity study of the Taiwan version of the Fukang Scale for the elderly in a community in Taipei City, including 400 elderly people in the community, including 142 who had fallen experience. The degree of reliability is 0.97, and the between-group reliability is 0.996.
Functional Fitness Test | one week
  Physical fitness is considered to be the comprehensive ability of the body to adapt to life and the environment; people with good physical fitness have good vitality and adaptability in daily life or work, physical activities or sports, and are not prone to fatigue or weakness; Ministry of Health and Welfare National Health Administration refers to the United States Scholars have designed functional fitness tests for the elderly over 60 years old, and developed domestic fitness tests to assess physical health. Topics include muscle strength and endurance, cardiorespiratory endurance, flexibility, agility, and homeostasis. Scholars in Taiwan conducted a reliability and validity study of the Taiwan version of the Fukang Scale for the elderly in a community in Taipei City, including 400 elderly people in the community, including 142 who had fallen experience. The degree of reliability is 0.97, and the between-group reliability is 0.996.
Functional Fitness Test | completed through training, usually two weeks
  Physical fitness is considered to be the comprehensive ability of the body to adapt to life and the environment; people with good physical fitness have good vitality and adaptability in daily life or work, physical activities or sports, and are not prone to fatigue or weakness; Ministry of Health and Welfare National Health Administration refers to the United States Scholars have designed functional fitness tests for the elderly over 60 years old, and developed domestic fitness tests to assess physical health. Topics include muscle strength and endurance, cardiorespiratory endurance, flexibility, agility, and homeostasis. Scholars in Taiwan conducted a reliability and validity study of the Taiwan version of the Fukang Scale for the elderly in a community in Taipei City, including 400 elderly people in the community, including 142 who had fallen experience. The degree of reliability is 0.97, and the between-group reliability is 0.996.
Tw-FROP-Com | first day
  Taiwan version of Falls Risk for Older People Community setting (Tw-FROP-Com) to evaluate risk factors associated with falls.in old adults. Falls in the old adults may not only cause physical and psychological harm, but also lead to death in severe cases, and may also increase medical costs.
  Taiwan introduced and fine-tuned the FROP-com scale designed by Russell et al. into the Taiwan version of the Fukang scale (TW-FROP-Com) to assess the risk of falls. The assessment contents include: fall experience, medication, medical conditions, whether Visual, somatosensory impairment, presence of foot or shoe problems, cognitive status, bladder control, nutritional status in the past three months and weight loss in the past year, environment, functional movements, activities of daily living (ADL) condition), walking balance, gait and activity; if the total score is more than 21 points, it is assessed as a high-risk group for falls.
Tw-FROP-Com | completed through training, usually two weeks
  Taiwan version of Falls Risk for Older People Community setting (Tw-FROP-Com) to evaluate risk factors associated with falls.in old adults. Falls in the old adults may not only cause physical and psychological harm, but also lead to death in severe cases, and may also increase medical costs.
  Taiwan introduced and fine-tuned the FROP-com scale designed by Russell et al. into the Taiwan version of the Fukang scale (TW-FROP-Com) to assess the risk of falls. The assessment contents include: fall experience, medication, medical conditions, whether Visual, somatosensory impairment, presence of foot or shoe problems, cognitive status, bladder control, nutritional status in the past three months and weight loss in the past year, environment, functional movements, activities of daily living (ADL) condition), walking balance, gait and activity; if the total score is more than 21 points, it is assessed as a high-risk group for falls.
Tw-FROP-Com | one week
  Taiwan version of Falls Risk for Older People Community setting (Tw-FROP-Com) to evaluate risk factors associated with falls.in old adults. Falls in the old adults may not only cause physical and psychological harm, but also lead to death in severe cases, and may also increase medical costs.
  Taiwan introduced and fine-tuned the FROP-com scale designed by Russell et al. into the Taiwan version of the Fukang scale (TW-FROP-Com) to assess the risk of falls. The assessment contents include: fall experience, medication, medical conditions, whether Visual, somatosensory impairment, presence of foot or shoe problems, cognitive status, bladder control, nutritional status in the past three months and weight loss in the past year, environment, functional movements, activities of daily living (ADL) condition), walking balance, gait and activity; if the total score is more than 21 points, it is assessed as a high-risk group for falls.

IPD SHARING:
Plan to Share IPD: No